CLINICAL TRIAL: NCT01729949
Title: A Randomized Placebo Controlled Trial to Test the Acute and Chronic Effects of Fruit Polyphenols on Postprandial Indices of Chronic Disease (PPF)
Brief Title: The Acute and Chronic Effects of Fruit Polyphenols on Chronic Disease (PPF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PPF 2012-073
Record Dates: First submitted 2012-11-08; First posted 2012-11-21 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Nutritional and Metabolic Disease; Overweight
Keywords: Nutrition; Polyphenols; Berries; Overweight; Lipid Panels
MeSH Terms: conditions — Metabolic Diseases; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment Beverage (Active Comparator): Strawberry powder and Blackcurrent extract
  Interventions: Dietary Supplement: Active Treatment Beverage
- Placebo Treatment Beverage (Placebo Comparator): Placebo Beverage
  Interventions: Dietary Supplement: Placebo Treatment Beverage

INTERVENTIONS:
Dietary Supplement: Active Treatment Beverage — Strawberry and Blackcurrent extract
  Other Names: Active Comparator
  Arms: Active Treatment Beverage
Dietary Supplement: Placebo Treatment Beverage — without active components
  Other Names: Placebo Comparator
  Arms: Placebo Treatment Beverage

SUMMARY:
1. The primary objective is to determine the effect of fruit polyphenols on postprandial lipoprotein triglyceride metabolism after consumption a standard high carbohydrate/fat breakfast meal with a beverage rich in fruit-derived polyphenols compared to energy and macro-/micro-nutrient matched control beverage (acute, Part 1).
2. Secondary objectives are: 1)to assess the effects of consuming daily for 8 weeks (chronic, Part 2) a beverage rich in fruit polyphenols compared to an energy and macro-/micro- nutrient matched control beverage on fasting glucose, insulin, lipids and markers of oxidative stress; and 2) to assess the effects of these beverages on meal-related changes in metabolic and oxidative stress measures after 8 weeks daily consumption.

DETAILED DESCRIPTION:
The study is a single-center, double-blinded, randomized, 2-part, 2-arm, 4-sequence, crossover study that incorporates both the acute and chronic evaluations of fruit polyphenols on metabolic indices and markers of oxidative stress.

A planned sample size of 30 overweight men and women will be recruited into the study. Subjects will be required to meet several inclusion and exclusion criteria, which will be assessed through online and clinic screening mechanisms, including questionnaires, blood analysis, and anthropometric measurements. Eligible subjects will be invited to participate in the study. Subjects will begin by completing a 7-day pre-study assessment of their usual dietary intake using 3-day food diary followed by washout of dietary polyphenols. Subjects will participate in 4, 6 h postprandial study days: 2 preceding the chronic intervention and 2 after 8 weeks each of active (fruit polyphenols) and placebo beverages. Subjects will be randomized on the first day of starting the acute and chronic study phases. Subjects will be asked to limit polyphenolic containing foods and beverages for 3 days prior to each 6 h postprandial study visit as well through the chronic dietary intervention. Subjects will be provided a standardized dinner meal pack on the day before each 6 h postprandial visit.

For each 6 h postprandial study visit, subjects will arrive fasted and follow procedures published by our lab previously. This includes: pre-study evaluation for compliance (fasting, dinner consumption, limited polyphenol intake) and readiness for study visit, catheter placement by registered nurse, fasting blood sample, consumption of high fat/carbohydrate meal accompanied by 1 of the two treatment beverages (active/fruit polyphenol or placebo beverage), subsequent blood sampling from catheter [ ~1 tablespoon (12ml)] at designated time points for 6 hours. Each postprandial study visit day will last approximately 7 hours and subjects will be required to remain at the Clinical Nutrition Research Center at the Illinois Institute of Technology main campus for the duration of the visit. The visit procedures are repeated twice ~ 1 week apart to accommodate subject testing with both beverages.

After completing both acute 6 h postprandial study visits, subjects will roll over to the chronic phase of the study and receive a 2nd randomization sequence for consuming the active or the placebo beverage daily for 8 weeks. Before crossing over to the alternative treatment beverage for another 8 weeks, subjects will have a 4-week break (wash out). Subjects will be counseled for a low polyphenolic diet throughout the study to consume the assigned beverage twice per day with lunch and evening meals (except during 4-week washout).

At the end of each week 8 treatment period, subjects will come to the research center for a 6 h postprandial study visit day: all procedures are identical on each postprandial study test visit with the exception that only the placebo beverage will be consumed with the breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking healthy overweight or class I obesity adult men and women
* Age 40-65yr
* Weight stable
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol.

Exclusion Criteria:

* Smokers or recent past smokers
* Men or women with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Diabetes
* Fasting blood glucose concentrations >125 mg/dL
* Fasting Total Cholesterol >250 mg/dL (6.47mmol/L)
* Fasting Triglycerides >250 mg/dL (2.82 mmol/L)
* Fasting LDL cholesterol >180 mg/dL (4.66 mmol/L)
* Uncontrolled blood pressure >140 mmHg/90 mmHg
* Documented vascular disease
* Cancer other than skin (non-melanoma) in previous 5 years
* Lactating and/or pregnant
* Taking medications or dietary supplements eg., antioxidant supplements, lipid lowering medication, blood pressure lowering medications.
* Recent blood donors (within 3 months)
* Vegans
* Substance (alcohol or drug) abuser (within the last 2 years)
* Participated in a chronic feeding or medication clinical trial in the last 3 months.
* Excessive coffee and tea consumers (> 4 cups/d)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2014-03-20 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Changes in Plasma Triglycerides Concentrations | Acute Postprandial (6 h) and chronic (8 week) fasting and postprandial (6 h)
  Changes in Plasma Triglyceride concentrations during the acute phases (from 0 to 6 hrs) and over the chronic phase, assessed by iAUC

SECONDARY OUTCOMES:
Changes in Plasma Lipid and Lipoprotein panels | Acute postprandial (6 h) and chronic (8 week) fasting and postprandial (6 h)
  Changes in Lipids (panel) and lipoprotein particle size/density by nuclear magnetic resonance (NMR)
Changes in insulin concentrations | Acute postprandial (6 h) and chronic (8 week) fasting and postprandial (6 h)
  Changes in Plasma insulin concentrations during the acute phases (from 0 to 6 hrs) and over the chronic phase, assessed by iAUC, total AUC, Cmax and TMax
Changes in LDL oxidation | Acute postprandial (6 h) and chronic (8 week) fasting and postprandial (6 h)
  Changes in Plasma OxLDL concentrations during the acute phases (from 0 to 6 hrs) and over the chronic phase, assessed by iAUC, total AUC, and Cmax
Changes in F2-isoprostane concentrations | Acute postprandial (6 h) and chronic (8 week) fasting and postprandial (6 h)
  Changes in Plasma F2-isoprostane concentrations during the acute phases (from 0 to 6 hrs) and over the chronic phases assessed by iAUC, total AUC, Cmax and TMax

OTHER OUTCOMES:
Changes in plasma glucose concentrations | Acute postprandial (6 h) and chronic (8 week) fasting and postprandial (6 h).
  Changes in Plasma glucose concentrations during the acute phases (from 0 to 6 hrs) and over the chronic phase, assessed by iAUC, total AUC, Cmax and TMax
Changes in polyphenol anthocyanin concentrations | Acute postprandial (6 h) and chronic (8 week) fasting and postprandial (6 h).
  Changes in Plasma polyphenol anthocyanin concentrations during the acute phases (from 0 to 6 hrs) and over the chronic phase, assessed by iAUC, total AUC, Cmax and TMax

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology; Indika Edirisinghe, Ph.D, Study Chair — Illinois Instutute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States